CLINICAL TRIAL: NCT01347255
Title: A Psoriasis Plaque Test Study With LEO 90100 Cutaneous Spray, Ointment, in Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: LEO 90100-01; 2011-000153-23
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2016-07

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Ointments; betamethasone-17,21-dipropionate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LEO 90100 cutaneous spray ointment (Experimental): LEO 90100 cutaneous spray, ointment, is a new product containing calcipotriol 50 mcg/g and betamethasone 0.5 mg/g (as dipropionate).
  Interventions: Drug: LEO90100 cutaneous spray, ointment
- LEO 90100 Cutaneous Spray, Ointment, Vehicle w. Betamethasone (Active Comparator): Vehicle cutaneous spray, ointment, with betamethasone 0.5 mg/g (as dipropionate)
  Interventions: Drug: LEO 90100 cutaneous spray, ointment, vehicle with betamethasone dipropionate
- LEO 90100 Cutaneous Spray, Ointment, Vehicle (Placebo Comparator): LEO 90100 vehicle served as a negative control for the two cutaneous spray ointments with active ingredients.
  Interventions: Drug: LEO 90100 cutaneous spray, ointment, vehicle
- Daivobet® Ointment (Active Comparator): Calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate)
  Interventions: Drug: Daivobet® ointment

INTERVENTIONS:
Drug: LEO90100 cutaneous spray, ointment — once daily application, 4 weeks
  Arms: LEO 90100 cutaneous spray ointment
Drug: LEO 90100 cutaneous spray, ointment, vehicle with betamethasone dipropionate — once daily application, 4 weeks
  Arms: LEO 90100 Cutaneous Spray, Ointment, Vehicle w. Betamethasone
Drug: LEO 90100 cutaneous spray, ointment, vehicle — once daily application, 4 weeks
  Arms: LEO 90100 Cutaneous Spray, Ointment, Vehicle
Drug: Daivobet® ointment — once daily application, 4 weeks
  Other Names: Taclonex® ointment
  Arms: Daivobet® Ointment

SUMMARY:
The purpose of the study is to evaluate the anti-psoriatic effect of LEO 90100 cutaneous spray ointment, using the psoriasis plaque test modified from the method developed by KJ Dumas and JR Scholtz.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects having signed and dated an informed consent
2. Age 18 years or above
3. Either sex
4. All skin types
5. Subjects with a diagnosis of psoriasis vulgaris with lesions located on arms, legs and/or trunk.

Exclusion Criteria:

1. Females who are pregnant, of child-bearing potential and who wish to become pregnant during the study, or who are breast feeding
2. Systemic treatment with biological therapies (marketed or not marketed) with a possible effect on psoriasis vulgaris within 4 weeks (etanercept), 2 months (adalimumab, alefacept, infliximab), 4 months (ustekinumab) or 4 weeks/5 half-lives (which-ever is longer)for experimental biological products prior to randomisation and during the study
3. Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, immunosuppressants) within the 4- week period prior to randomisation and during the study
4. Use of phototherapy within the following time periods prior to randomisation and during the study:

   * PUVA or Grenz ray therapy (4 weeks)
   * UVB (2 weeks)
5. Subjects using one of the following topical drugs within 4 weeks prior to randomisation and during the study:

   * Potent or very potent (WHO group III-IV) corticosteroids
6. Subjects using one of the following topical drugs for the treatment of psoriasis within 2 weeks prior to randomisation and during the study:

   * WHO group I-II corticosteroids (except if used for treatment of scalp and/or facial psoriasis)
   * Topical retinoids
   * Vitamin D analogues
   * Topical immunomodulators (e.g. calcineurin inhibitors)
   * Anthracen derivatives
   * Tar
   * Salicylic acid
7. Subjects using emollients on the target plaques within one week before randomisation and during the study
8. Initiation of, or expected changes in concomitant medication that may affect psoriasis vulgaris (e.g., beta blockers, anti-malaria drugs, lithium and ACE inhibitors) within 2 weeks prior to randomisation and during the study
9. Subjects with current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis
10. Subjects with known/suspected disorders of calcium metabolism associated with hypercalcemia within the last 10 years, based on medical history
11. Subjects with any of the following conditions present on the test area: viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections and atrophic skin
12. Subjects with skin manifestations in relation to syphilis or tuberculosis, rosacea, perioral dermatitis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, acne rosacea, ulcers and wounds within the plaque test areas
13. History of any severe disease or serious current condition (based on subject interview and/or results of screening physical examination) which, in the opinion of the Investigator, would put the subject at risk by participating in the study or would interfere significantly with the evaluation of study results or the study course (e.g. cancer, severe cardiopathy, severe renal insufficiency, severe hepatic insufficiency)
14. Subjects who have received treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within the 4 week period prior to randomisation or longer, if the class of the substance requires a longer washout as defined above (e.g., biological treatments)
15. Subjects with current participation in any other interventional clinical trial, based on interview of the subject
16. Subjects with known or suspected hypersensitivity to component(s) of the investigational products
17. Subjects with any concomitant medical or dermatological disorder(s) which might preclude accurate evaluation of the psoriasis
18. Subjects foreseeing an intensive solar exposure during the study (UV radiation, etc.) or having been exposed within two weeks preceding the screening visit
19. Subjects impossible to contact in case of emergency
20. Subjects who are known or, in the opinion of the investigator, are unlikely to comply with the Clinical Study Protocol (e.g. alcoholism, drug dependency or psychotic state)
21. Subjects who are in an exclusion period in the National Biomedical Research Register of the French Ministry of Health at randomisation
22. Subjects under guardianship, hospitalized in a public or private institution, for a reason other than the research or subject deprived of freedom
23. Subjects previously randomised in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Queille-Roussel, MD, Principal Investigator — Centre de Pharmacologie Clinique Appliquée à la Dermatologie (CPCAD), Hôpital l'Archet 2, 06202 Nice Cedex 3, France
Locations (1):
- Centre de Pharmacologie Clinique Appliquée à la Dermatologie (CPCAD), Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Queille-Roussel C, Olesen M, Villumsen J, Lacour JP. Efficacy of an innovative aerosol foam formulation of fixed combination calcipotriol plus betamethasone dipropionate in patients with psoriasis vulgaris. Clin Drug Investig. 2015 Apr;35(4):239-45. doi: 10.1007/s40261-015-0269-7. PMID 25708531
- [Result] Queille-Roussel C, Olesen M, Villumsen J, Lacour JP. Antipsoriatic effect of a novel aerosol foam formulation of the fixed combination calcipotriene plus betamethasone dipropionate in patients with psoriasis, using a modified psoriasis plaque test. Semin Cutan Med Surg. 2015;34 S1:PA-10.
- [Result] Hollesen Basse L, Olesen M, Lacour J, Queille-Roussel C. Enhanced in vitro skin penetration and antipsoriatic effect of fixed combination calcipotriol plus betamethasone dipropionate in an innovative foam vehicle. J Invest Dermatol. 2014;134:S33(abst 192).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 12-MAY-2011 Last Subject Last Visit: 20-JUN-2011
Pre-assignment Details: The study was conducted with 3 successive individual phases:
  * Screening Phase (washout if applic.). A medical examination was performed at screening which took place 1-21 days before the start of the treatment phase (Day 1).
  * Treatment Phase (All patients (N=24) received all investigational medicinal products)
  * Follow-up Phase (if applic.)
Groups:
- All Study Participants: All subjects received all four treatments:
  1. LEO 90100 cutaneous spray, ointment, is a new product containing calcipotriol 50 mcg/g and betamethasone 0.5 mg/g (as dipropionate)
  2. LEO 90100 cutaneous spray, ointment, vehicle w. betamethasone. Vehicle cutaneous spray, ointment, with betamethasone 0.5 mg/g (as dipropionate)
  3. LEO 90100 cutaneous spray, ointment, vehicle. Served as a negative control for the two cutaneous spray ointments with active ingredients
  4. Daivobet® ointment. Calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate)
  Four test sites of approximately 5 cm2 were selected on predetermined psoriasis lesions (target plaques), delimited with a disposable circular device and mapped on a drawn figure.
  The distance between two test sites was at least 2 cm. The products were applied on the four test sites (according to random assignment to specific test sites selected on the psoriasis plaque) once daily 6 days a week (except Sundays) for 4 weeks.
Period: Overall Study
Arm/Group | All Study Participants
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intra-individual baseline analysis population
Groups:
- LEO 90100 Cutaneous Spray, Ointment: Intra-Individual baseline analysis population, all treated with the following four products:
  1. LEO 90100 cutaneous spray, ointment: once daily application, 4 weeks (6 days a week)
  2. LEO 90100 cutaneous spray, ointment, vehicle with betamethasone dipropionate: once daily application, 4 weeks (6 days a week)
  3. LEO 90100 cutaneous spray, ointment, vehicle: once daily application, 4 weeks (6 days a week)
  4. Daivobet® ointment: once daily application, 4 weeks (6 days a week)
Arm/Group | LEO 90100 Cutaneous Spray, Ointment
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Total Clinical Score (TCS) of Clinical Signs (Sum of Erythema, Scaling and Infiltration) at End of Treatment Compared to Baseline
Description: TCS range from 0 (all signs absent) to 9 (all signs severe).
Time Frame: Day 1 (Baseline)/Day 29
Population: Intra-individual analysis population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- LEO 90100 Cutaneous Spray, Ointment: LEO 90100 cutaneous spray, ointment, is a new product containing calcipotriol 50 mcg/g and betamethasone 0.5 mg/g (as dipropionate).
Arm/Group | LEO 90100 Cutaneous Spray, Ointment | LEO 90100 Cutaneous Spray, Ointment, Vehicle w. Betamethasone | LEO 90100 Cutaneous Spray, Ointment, Vehicle | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24
Scores on a scale | -6.00 (1.27) | -4.96 (1.85) | -1.88 (1.12) | -5.25 (1.78)

2. Secondary Outcome: Change in Clinical Sign Scores
Description: Absolute change in score of each clinical sign (erythema, scaling, infiltration) at end of treatment (Day 29) and at individual visits (Days 4, 8, 11, 15, 18, 22, and 25) compared to Baseline.
  The investigator assessed the severity of the clinical signs erythema, scaling, and infiltration for each test site by using a 7-point scale (range 0 (no evidence) to 3 (severe)).
  Negative changes in mean score represent improvement.
Time Frame: Baseline and Days 4, 8, 11, 15, 18, 22, 25, and 29 (End of Treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEO 90100 Cutaneous Spray, Ointment | LEO 90100 Cutaneous Spray, Ointment, Vehicle w. Betamethasone | LEO 90100 Cutaneous Spray, Ointment, Vehicle | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale
  Erythema (Day 29) | -1.75 (0.71) | -1.44 (0.78) | -0.56 (0.47) | -1.50 (0.66)
  Scaling (Day 29) | -2.13 (0.47) | -2.02 (0.58) | -0.90 (0.47) | -2.02 (0.56)
  Infiltration (Day 29) | -2.13 (0.45) | -1.50 (0.77) | -0.42 (0.43) | -1.73 (0.82)
  Erythema (Day 4) | -0.33 (0.32) | -0.33 (0.32) | -0.19 (0.25) | -0.33 (0.32)
  Scaling (Day 4) | -0.17 (0.35) | -0.31 (0.36) | -0.19 (0.25) | -0.23 (0.36)
  Infiltration (Day 4) | -0.13 (0.30) | -0.13 (0.27) | -0.08 (0.19) | -0.17 (0.28)
  Erythema (Day 8) | -0.73 (0.42) | -0.60 (0.42) | -0.13 (0.37) | -0.67 (0.43)
  Scaling (Day 8) | -0.75 (0.66) | -0.81 (0.59) | -0.21 (0.44) | -0.73 (0.64)
  Infiltration (Day 8) | -0.60 (0.39) | -0.42 (0.43) | -0.08 (0.41) | -0.56 (0.54)
  Erythema (Day 11) | -1.08 (0.46) | -0.75 (0.42) | -0.29 (0.39) | -0.83 (0.52)
  Scaling (Day 11) | -1.29 (0.67) | -1.06 (0.70) | -0.46 (0.49) | -1.23 (0.68)
  Infiltration (Day 11) | -1.00 (0.47) | -0.58 (0.52) | -0.23 (0.44) | -0.90 (0.55)
  Erythema (Day 15) | -1.29 (0.41) | -1.06 (0.52) | -0.33 (0.43) | -1.04 (0.55)
  Scaling (Day 15) | -1.65 (0.63) | -1.40 (0.59) | -0.46 (0.41) | -1.40 (0.61)
  Infiltration (Day 15) | -1.31 (0.44) | -0.85 (0.52) | -0.23 (0.44) | -1.06 (0.68)
  Erythema (Day 18) | -1.37 (0.43) | -1.20 (0.62) | -0.35 (0.41) | -1.35 (0.41)
  Scaling (Day 18) | -1.87 (0.57) | -1.52 (0.67) | -0.67 (0.44) | -1.74 (0.64)
  Infiltration (Day 18) | -1.61 (0.54) | -1.11 (0.62) | -0.30 (0.45) | -1.43 (0.70)
  Erythema (Day 22) | -1.79 (0.55) | -1.29 (0.46) | -0.52 (0.43) | -1.44 (0.58)
  Scaling (Day 22) | -2.06 (0.54) | -1.73 (0.64) | -0.67 (0.48) | -1.81 (0.55)
  Infiltration (Day 22) | -1.85 (0.50) | -1.35 (0.67) | -0.38 (0.42) | -1.50 (0.69)
  Erythema (Day 25) | -1.79 (0.53) | -1.44 (0.68) | -0.56 (0.43) | -1.56 (0.68)
  Scaling (Day 25) | -2.15 (0.50) | -1.98 (0.60) | -0.85 (0.38) | -1.98 (0.56)
  Infiltration (Day 25) | -2.10 (0.49) | -1.52 (0.67) | -0.44 (0.37) | -1.67 (0.72)

3. Secondary Outcome: Changes in Total Clinical Score (TCS) by Visit
Description: Change in Total Clinical Score (TCS; range from 0 (all signs absent) to 9 (all signs severe)) at individual visits (Days 4, 8, 11, 15, 22, and 25) compared to baseline.
Time Frame: Baseline and Days 4, 8, 11, 15, 18, 22, 25
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LEO 90100 Cutaneous Spray, Ointment | LEO 90100 Cutaneous Spray, Ointment, Vehicle w. Betamethasone | LEO 90100 Cutaneous Spray, Ointment, Vehicle | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24
Scores on a scale
  Day 4 | -0.63 (0.65) | -0.77 (0.71) | -0.46 (0.36) | -0.73 (0.71)
  Day 8 | -2.08 (1.17) | -1.83 (1.03) | -0.42 (0.83) | -1.96 (1.28)
  Day 11 | -3.38 (1.17) | -2.40 (1.38) | -0.98 (0.87) | -2.96 (1.41)
  Day 15 | -4.25 (1.07) | -3.31 (1.31) | -1.02 (0.94) | -3.50 (1.54)
  Day 18 | -4.85 (1.17) | -3.83 (1.66) | -1.33 (1.00) | -4.52 (1.42)
  Day 22 | -5.71 (1.17) | -4.38 (1.49) | -1.56 (1.08) | -4.75 (1.52)
  Day 25 | -6.04 (1.15) | -4.94 (1.68) | -1.85 (0.88) | -5.21 (1.68)

4. Secondary Outcome: Change From Baseline in Echo-poor Band Thickness at End of Treatment
Description: Change in echo-poor band thickness from baseline to end of treatment, measured by ultrasound
Time Frame: Baseline and Day 29
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | LEO 90100 Cutaneous Spray, Ointment | LEO 90100 Cutaneous Spray, Ointment, Vehicle w. Betamethasone | LEO 90100 Cutaneous Spray, Ointment, Vehicle | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24
millimetres | -0.57 (0.21) | -0.45 (0.25) | -0.12 (0.20) | -0.46 (0.21)

5. Secondary Outcome: Changes in Total Skin Thickness
Description: Change in total skin thickness measured by ultrasound at end of treatment (Day 29) and individual visits (Days 8, 15, and 22) compared to baseline
Time Frame: Baseline and Days 8, 15, 22, and 29.
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | LEO 90100 Cutaneous Spray, Ointment | LEO 90100 Cutaneous Spray, Ointment, Vehicle w. Betamethasone | LEO 90100 Cutaneous Spray, Ointment, Vehicle | Daivobet® Ointment
Number analyzed (Participants) | 24 | 24 | 24 | 24
millimetres
  Day 29 | -0.81 (0.41) | -0.66 (0.42) | -0.23 (0.30) | -0.62 (0.37)
  Day 8 | -0.37 (0.31) | -0.28 (0.19) | -0.07 (0.21) | -0.33 (0.24)
  Day 15 | -0.57 (0.38) | -0.40 (0.29) | -0.12 (0.23) | -0.49 (0.26)
  Day 22 | -0.68 (0.40) | -0.59 (0.35) | -0.18 (0.25) | -0.59 (0.33)

ADVERSE EVENTS:
Groups:
- LEO 90100 Cutaneous Spray, Ointment: Intra-Individual baseline analysis population, all treated with the following four products:
  1. LEO 90100 cutaneous spray, ointment: once daily application, 4weeks
  2. LEO 90100 cutaneous spray, ointment, vehicle with betamethasone dipropionate: once daily application, 4 weeks
  3. LEO 90100 cutaneous spray, ointment, vehicle: once daily application, 4weeks
  4. Daivobet® ointment: once daily application, 4weeks
Arm/Group | LEO 90100 Cutaneous Spray, Ointment
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 10/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 Cutaneous Spray, Ointment (N=24)
Toothache (Gastrointestinal disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.